CLINICAL TRIAL: NCT01241981
Title: Digital Breast Tomosynthesis (DBT): Sensitivity for Cancer and Accuracy in Assessing Extent of Malignant Disease in Symptomatic Women Below 60 With Clinical or Ultrasound Signs Compatible With Malignancy
Brief Title: Digital Breast Tomosynthesis in Younger Symptomatic Women
Status: Completed | Type: Observational
Sponsor: NHS Tayside (Other Government)
Collaborators: University of Dundee (Other)
Responsible Party: Principal Investigator, Andy Evans, Professor of Breast Imaging, NHS Tayside
Other Study IDs: 2010ON15
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; Digital; Mammography; Tomosynthesis
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Digital Breast Tomosynthesis: Digital Breast Tomosynthesis

SUMMARY:
This study will examine a new imaging technique called digital breast tomosynthesis (DBT) compared to standard mammography in women under 60 presenting with signs of breast cancer. The reason that we need to do this study is that standard mammography fails to detect the cancer in approximately 20% of these women because younger women have denser breast tissue. We hope that DBT will be more sensitive in detecting breast cancer than standard mammography.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Under 60 years old
* Clinical or ultrasound suspicion of breast cancer

Exclusion Criteria:

* Unable to give informed consent
* Male
* Obvious advanced breast cancer
* Obvious medical problems meaning surgery would not be an option

Max Age: 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women under 60 years of age with clinical or ultrasound suspicion of breast cancer
Sampling Method: Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2011-03; Primary Completion 2016-12-21 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity of DBT for breast cancer, compared with FFDM | Two years

SECONDARY OUTCOMES:
Accuracy of DBT compared with FFDM in assessment of tumour extent | Two years
Relative accuracy of DBT and FFDM by breast density | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Evans, FRCR, Principal Investigator — University of Dundee, NHS Tayside
Locations (1):
- NHS Tayside, Ninewells Hospital & Medical School, Dundee, Tayside, United Kingdom